CLINICAL TRIAL: NCT03457532
Title: An Open-label, Multicenter, Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics Characters, and Preliminary Efficacy of SCC244 in Patients with Advanced MET Alterations Solid Tumors
Brief Title: A Phase I Study of SCC244 in Patients with Advanced MET Alterations Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haihe Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCC244-104
Record Dates: First submitted 2018-02-09; First posted 2018-03-07 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumor
Keywords: Safety, Tolerability, Pharmacokinetics, Anti-tumor Activity
MeSH Terms: interventions — glumetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose escalation study of Gumarontinib (Experimental): To determine the maximum tolerated dose (MTD) of Gumarontinib
  Interventions: Drug: Gumarontinib Tablets

INTERVENTIONS:
Drug: Gumarontinib Tablets — 25mg; 50mg; 100mg; 200mg; 400mg; 600mg BID or QD(Decided by SMC accroding to the safty and PK data)
  Other Names: SCC244

SUMMARY:
This is a Phase 1a/1b multi-center and open label study to evaluate the safety, tolorability, pharmacokinetics and priliminary efficacy of SCC244 in advanced solid tumors patients with c-MET alteration

DETAILED DESCRIPTION:
This is a phase I study, its purpose to evaluate the safety and tolerability and to determine the maximum tolerated dose (MTD)/ biologically effective dose (BED) and the recommended phase II dose (RP2D) of SCC244 monotherapy in patients with advanced MET alterations solid tumors;

ELIGIBILITY:
Main Inclusion:

1. Fully understand the study and signed the informed consent must be obtained prior to any screening procedures.
2. Adults are more than 18 years old at the time of informed consent.
3. Life expectancy is more than 12 weeks by the Investigator's discretion.
4. For phase Ia study and cohort 1 in phase Ib study: Patients with histologically or cytologically confirmed locally advanced or metastatic solid tumors who failed the standard treatment or with no standard treatment available. For cohort 2 in phase Ib study: a) Patients with stage IIIb or IIIc NSCLC who are not candidates for definitive surgical resection or concurrent chemoradiation or patients with stage IV NSCLC (including PSC) confirmed histologically or cytologically. b) Patients who received is less than 2 lines of prior anti-tumor systemic therapy and had not previously used MET inhibitors. c) Participants with advanced/metastatic NSCLC must be unsuitable for chemotherapy or refused chemotherapy after fully informed or have failed one or two prior lines of systemic therapy
5. Patients with MET alteration：1) MET amplification; 2) MET over-expression; 3）MET axon 14 skipping mutation or 4) MET fusion;
6. At least 1 measurable target lesion according to RECIST 1.1;
7. ECOG performance status of 0-1;
8. Patients with HCC must be satisfied with liver function of Child Pugh Class A;
9. Patients must have adequate organ function;
10. International normalized ratio (INR) is less than 1.5 or activated partial thromboplastin time (aPTT) is less than 1.5 x ULN;
11. Patients must have recovered from all toxicities related to prior anticancer therapies to grade is less than 1 (CTCAE v 4.03) with the exception of alopecia and grade 2 prior neuropathy;
12. Patients who are willing and able to receive scheduled visits, treatment plan, laboratory tests and other required study procedures;
13. Males and females of child-bearing potential must agree to use highly effective methods of contraception during dosing and for 6 months after stopping treatment. Males with pregnancy or nursing partner must adopt double barrier contraception to prevent sperm from affecting the fetus or child;
14. Female patients can only participate in this study;

Main Exlcusion:

1. Known druggable molecular alterations such as EGFR mutation, ALK rearrangement, ROS1 rearrangement, BRAF mutation, or NTRK fusion which might be a candidate for alternative targeted therapies as applicable per local regulations and treatment guidelines;
2. Pregnant or nursing women;
3. Previous anti-cancer therapies must be discontinued 4 weeks or 5×half-life of the agent before first dose of SCC244. If previous treatment is a monoclonal antibody, the treatment must be discontinued 2 weeks or 5×half-life of the agent before first dose of SCC244. Traditional Chinese medicine with anti-tumor indications must be discontinued 2 weeks before first dose of SCC244.
4. Patients receiving treatment with strong inhibitors or strong inducers of CYP3A4
5. Any major surgery or significant traumatic injury within 4 weeks prior to the first investigational product administration.
6. Radical radiotherapy within 4 weeks prior to the first investigational product administration., or locally palliative radiotherapy within 2 weeks prior to the first investigational product administration.
7. Other prior or concomitant primary malignancies.
8. Patients with clinically significant cardiovascular system disease
9. History of stroke within 6 months prior to screening.
10. Requiring total brain radiotherapy for control of brain metastases. Patients with symptomatic brain metastases who are expected to receive local brain treatment during protocol treatment will also be not eligible for the study. If patients require steroids for brain metastases, the daily dose should not exceed 10 mg of dexamethasone or equivalent of other steroids.
11. Unable to swallow oral medicine, active digestive system diseases, or major digestive tract surgery that may affect the administration and absorption of SCC244 according to the judgment of the investigator.
12. Any clinically significant disease or condition that may affect compliance to the protocol.
13. Patients with positive HBsAg and serum HBV DNA is less than 1000 copies/ml or 200 IU/ml who are clinically confirmed to be inactive infections will be eligible for the study. Prophylactic anti-HBV medication is acceptable. However, patients with positive test for anti-HCV antibody or HCV RNA should be excluded.
14. Known HIV infection.
15. Unable to discontinue some specific medications;
16. History of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis requiring steroid therapy, or any evidence of clinically active ILD;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2017-12-16 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
DLT(Dose limit toxity) | 35 days
  To evaluate the DLT in patients with advanced solid tumor
MTD(Max tolerance does) | 35 days
  To evaluate the MTD in patients with advanced solid tumor
BED(Biological effective dose) | 35 days
  To evaluate the BED in patients with advanced solid tumor
objective response rate (ORR) | 8 weeks
  To evaluate the ORR in patients with advanced solid tumor in Ib

CONTACTS AND LOCATIONS:
Overall Officials: Fugen Li, Study Chair — Haihe Biopharma Co., Ltd.
Locations (1):
- Shanghai East hospital, Shanghai, China

REFERENCES:
- [Derived] Yu Y, Dong W, Shi Y, Wu R, Yu Q, Ye F, Zhou C, Dong X, Li X, Li Y, Li Z, Wu L, Pan Y, Shen H, Wu D, Xu Z, Wu J, Xu N, Qin Y, Zang A, Zhang J, Zhou J, Zhang X, Zhao Y, Li F, Wang H, Liu Q, Han Z, Li J, Lu S. A pooled analysis of clinical outcome in driver-gene negative non-small cell lung cancer patients with MET overexpression treated with gumarontinib. Ther Adv Med Oncol. 2024 Jul 31;16:17588359241264730. doi: 10.1177/17588359241264730. eCollection 2024. PMID 39091606